CLINICAL TRIAL: NCT00910559
Title: Phenotypic and Genetic Factors in Autism Spectrum Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Christopher Walsh, Professor of Genetics and Pediatrics, Harvard Medical School, Boston Children's Hospital
Other Study IDs: 04-05-075; R01MH085143 (NIH); R01MH083565 (NIH)
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorder; Autism; Asperger Syndrome; Pervasive Developmental Disorders- Not Otherwise Specified
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to collect phenotypic (observable characteristics) and genetic information about individuals with Autism Spectrum Disorders (ASDs) and their families.

DETAILED DESCRIPTION:
Participation in this research study involves two research visits, at least one of which is at Children's Hospital Boston. The first visit lasts about 4-6 hours. On this visit, the child will work with a research assistant on a few different cognitive assessments while one or both parents answer interview questionnaires about the child's development, along with other family history information. The second visit at the hospital lasts about 2 and a half hours and involves medical history and family history questionnaires, as well as height, weight, and head circumference measurements and a blood draw from each family member. In addition, digital photographs will be taken of each family member and a 3-D picture of the child's face will be taken. Shortly after the visits, participants will receive a research report of our observations. These results include cognitive, behavioral, developmental, and social findings. The total time commitment for the study is 6 to 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder or suspected diagnosis based on clinical genetic test results (e.g., variant diagnosed via chromosomal microarray)
* Age ≥ 18 months

Exclusion Criteria:

* Presence of a metabolic disorder
* Acquired developmental disability (e.g., birth asphyxia, trauma-related injury, meningitis, etc.) or cerebral palsy

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with ASDs and their parents and/or siblings
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2008-07; Primary Completion 2028-01 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
genotype-phenotype correlation | enrollment and sample analysis

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Walsh, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data is available through National Database for Autism Research (NDAR) and database of Genotypes and Phenotypes (dbGaP).